CLINICAL TRIAL: NCT06908135
Title: Effects of an Independent Walking Program With Walking Poles in People With Parkinson Disease
Acronym: ActivatePD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Northwest University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-032
Record Dates: First submitted 2025-03-12; First posted 2025-04-03 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: walking; physical activity; gait; arm swing; Nordic walking
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single center, two arm, pre-test post-test parallel design with 2 cohorts of participants.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Walking Poles (Experimental): Participants who will be using walking poles
  Interventions: Behavioral: Independent walking program using walking poles
- No Walking Poles (Active Comparator): Participants who will not be using walking poles
  Interventions: Behavioral: Independent walking program without walking poles

INTERVENTIONS:
Behavioral: Independent walking program using walking poles — Participants will independently walk at least 3 times a week for 8 weeks using walking poles
  Arms: Walking Poles
Behavioral: Independent walking program without walking poles — Participants will independently walk at least 3 times a week for 8 weeks without walking poles
  Arms: No Walking Poles

SUMMARY:
* Study Purpose: The purpose of the study is to compare changes in activity levels and walking in people with Parkinson disease after an 8-week independent walking program with or without using walking poles.
* Major parts of the Study:

Before the walking program: You will wear an activity sensor on your upper leg for one week to track activity levels. Measurements will be taken of you while you are walking. If you are placed in the walking pole group, you will be trained on how to use walking poles.

Independent walking program: You will be asked to walk at least 3 times each week for 8 weeks and keep a log of your walking. If you are in the walking pole group, you will walk with the poles.

After the walking program: Your walking measurements will be collected as before the walking program. You will wear an activity sensor for one week.

DETAILED DESCRIPTION:
The study will be comprised of a pre-visit distribution of the consent form with an opportunity to ask questions during a phone conversation, and 4 in-person visits in total: (1) consent signature, written outcomes, and activity sensor placement, (2) activity sensor collection and initial baseline testing, (3) post-intervention testing, written outcomes, and activity sensor placement, and (4) activity sensor collection. Each participant will be assigned a study ID number consisting of a root '0203' appended by the participant number (ie, '01', '02', etc), assigned in order of initial testing. (e.g., the first participant ID will be 020301).

Prior to Visit 1, the consent form will be emailed (preferred) or mailed to the potential participant for review. If the potential participant wishes, they will be contacted by phone by the PI or a co-Investigator and the study will be explained, inclusion and exclusion criteria will be reviewed and recorded on the Eligibility Form (see attached), and the potential participant will be given the opportunity to ask questions regarding the study.

Visit 1 will include answering any outstanding questions and obtaining a signature indicating informed consent, obtaining participant demographics and written outcome measures, application of the activity sensor, and giving the participant the Medical Clearance Form.

* Participants will be asked to verbalize understanding and will be asked if they have any questions about the study before being asked to sign the Consent Form.
* Participant demographics will include age, weight, height, gender, years since diagnosis, Hoehn & Yahr stage, daily levodopa intake and the following questions: "Are you comfortable using walking/hiking poles?" and "How many days per week do you participate in intentional exercise?" These data will be recorded on the Outcome Measures Spreadsheet (see attached).
* Written outcome measure will include: Trail Making Test Parts A and B, Activities Specific Balance Confidence Scale (ABC Scale), Parkinson Disease Questionnaire Shortened Form (PDQ-8)
* An activPAL™ sensor will be secured to the anterior thigh of their less-involved side (if applicable). Medical tape or transparent film dressing will be used to secure the sensor. Showering with the sensor on is permitted. If the participant may submerge in water (i.e., bathing or swimming) during the week or if the participant prefers, transparent film dressing will be used to attach and waterproof the sensor.
* The Medical Clearance Form (see attached) will be provided to the participant for completion by their provider. The Medical Clearance Form must be returned to the PI prior to the walking program portion of the study.

Visit 2 will include baseline assessments and study group assignment.

* The activPAL™ sensor and Medical Clearance Form will be collected.
* Outcome measures will include: 10-meter walk test for gait speed and characteristics without walking poles on the Zeno™ Walkway, 4-square step test without walking poles on the Zeno™ Walkway, and the 6-minute walk test with the portable Zeno™ Walkway in the test course loop, Ultium MyoMOTION™ sensors strapped on each wrist, and 2 to 4 Ultium MyoMUSCLE™ EMG sensors affixed to the trunk. Gait characteristics will concurrently be collected with the above tests performed on the respective Zeno™ Walkway. MyoMOTION™ sensors will collect arm swing data and MyoMUSCLE™ sensors will collect muscle activation data. (see Section 5.5 for details)

  * The manually collected data will be recorded on the Outcome Measures spreadsheet.
  * Gait characteristic data is collected with the Zeno™ Walkway software (PKMAS).
  * Arm swing data is collected with the Ultium MyoMOTION™ software (MyoRESEARCH™ 4).
  * Trunk muscle activation data is collected with the Ultium MyoMUSCLE™ software (MyoRESEARCH™ 4).
* Within 2 days of the baseline assessment, participants will participate in a group training on the use of walking poles, including fitting and practice with the poles. The class will last no more than 60 minutes, although the PI/instructor will provide training for as long as participants desire.

  * Immediately before training, participants will perform the 10-meter walk test without poles on the Zeno™Walkway.
  * Immediately after training, the participants will repeat the 10-meter walk test with and without walking poles on the Zeno™ Walkway.
  * After training and the gait assessment data are collected, the study group allocation will be revealed to each participant by a study member not involved in the assessment data collection.
  * Participants randomized into the walking pole group will be provided with the poles for home use and asked to use the poles during all walking for exercise during the study period. Pole use will not be restricted outside of the walking program.

Walking program period:

* All participants (intervention and control) will be asked to participate in at least 3 days of intentional walking exercise for the subsequent 8 weeks. Each participant will be given a log (see attached) to record their walking frequency and duration, rating of perceived exertion (RPE), notes, and any adverse events. Participants will be educated on the RPE scale and provided with a laminated RPE scale (see attached). All participants will be instructed to contact the PI via phone or email if an adverse event occurs. Events are defined as "Illness, injury, or falls" and contact information is provided on each page of the log.
* Participants will be contacted by a study member (see Check-in Script) by email (preferred) or phone (if participant does not use email or does not respond to email within 48 hours) at the end of weeks 1, 2, 4 and 6.

Visit 3 occurs at the conclusion of the 8-week walking program.

* Walking logs will be collected.
* Outcome measures will be collected, including: Trail Making Test Parts A and B, Activities Specific Balance Confidence Scale (ABC Scale), Parkinson Disease Questionnaire Shortened Form (PDQ-8), 10-meter walk test for gait speed and characteristics with and without walking poles on the Zeno™ Walkway, 4-square step test with and without walking poles on the Zeno™ Walkway, and the 6-minute walk test with the portable Zeno™ Walkway in the test course loop, Ultium MyoMOTION™ sensors strapped on each wrist, and 2 to 4 Ultium MyoMUSCLE™ EMG sensors affixed to the trunk. Gait characteristics will concurrently be collected with the above tests performed on the respective Zeno™ Walkway. MyoMOTION™ sensors will collect arm swing symmetry and amplitude and MyoMUSCLE™ sensors will collect muscle activation data.
* An ActivPAL™ sensor will be secured to the anterior thigh of the participants' less-involved side (if applicable). Medical tape or transparent film dressing will be used to secure the sensor. Showering with the sensor on is permitted. If the participant may submerge in water (i.e., bathing or swimming) during the week or if the participant prefers, transparent film dressing will be used to attach and waterproof the sensor.

Visit 4

* The ActivPAL™ sensor will be collected.
* Participants in the control group will be given a pair of walking poles for personal use.

At 3 months post-completion, participants will be contacted by email or phone to complete an ABC Scale and PDQ-8 questionnaire. Participants will be asked to estimate how many times in the past 2 weeks they went for an intentional walk and if they used the walking poles for those walks.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of Parkinson disease,
2. ability to walk independently with or without a cane,
3. receive medical clearance to participate in an independent walking,
4. English or Spanish language proficiency at 8th grade level.

Exclusion Criteria:

1. diagnosis of any neurological disease other than PD (including but not limited to stroke, dementia, and multiple sclerosis; mild cognitive impairment is not excluded),
2. use of walking poles during walking for exercise more than 4 times during the last year (hiking with poles permitted),
3. weight of more than 320 lb or height more than 6'4",
4. allergy to medical-grade adhesive,
5. unable to participate in walking for more than 5 consecutive days during the study period (ie, traveling, scheduled surgery),
6. a change in Parkinson medication that affects Levodopa levels (including additions, removals, or changes in dosage) during the study period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Gait Characteristic - gait speed | Prior to initiation of 8 week walking program and immediately upon completion.
  Gait characteristics collected on Zenomat walkway, including gait speed (m/s)
Gait Characteristic - step length | Prior to initiation of 8 week walking program and immediately upon completion.
  Gait characteristics collected on Zenomat walkway, including step length (m)
Gait Characteristic - step symmetry | Prior to initiation of 8 week walking program and immediately upon completion.
  Gait characteristics collected on Zenomat walkway, including step symmetry (symmetry index, %)
Gait Characteristic - gait variability | Prior to initiation of 8 week walking program and immediately upon completion.
  Gait characteristics collected on Zenomat walkway, including gait variability (enhanced gait variability index)

SECONDARY OUTCOMES:
Physical Activity | Upon enrollment for 1 week, followed by 8 week independent walking program with no activity monitoring, then upon walking program completion for 1 week.
  Measurement of time spent in each activity each day - seated, walking, standing, and lying obtained using the ActivPAL sensors. (time - hours:minutes)
Physical Activity - daily steps | Upon enrollment for 1 week, followed by 8 week independent walking program with no activity monitoring, then upon walking program completion for 1 week.
  Measurement of daily steps obtained using the ActivPAL sensors. (# counted)
Physical Activity - daily sit to stands | Upon enrollment for 1 week, followed by 8 week independent walking program with no activity monitoring, then upon walking program completion for 1 week.
  Measurement of count of sit to stands obtained using the ActivPAL sensors. (# counted)
Physical Activity - activity score | Upon enrollment for 1 week, followed by 8 week independent walking program with no activity monitoring, then upon walking program completion for 1 week.
  Measurement of activity score in metabolic equivalents (METs) obtained using the ActivPAL sensors. (METs)
Four Square Step Test | Prior to initiation of 8 week walking program and immediately upon completion.
  Four Square Step Test measurements taken on Zenomat and are a test of dynamic balance and coordination that assesses the participant's ability to step over objects forward, sideways, and backwards. Measurements include test completion time and step characteristics.
Arm swing | Prior to initiation of 8 week walking program and immediately upon completion.
  Arm swing data collected via inertial measurement unit (IMU) sensors on arms to measure angle and excursion; collected concurrently with gait data.
Cervical and lumbar extensor muscle activation | Prior to initiation of 8 week walking program and immediately upon completion.
  Collected via electromyography (EMG) sensors affixed over cervical and lumbar spinal extensors; collected concurrently with gait data.
Activity-specific Balance Confidence Scale | Prior to initiation of 8 week walking program and immediately upon completion
  Self-administered questionnaire that reflects the participant's confidence in their ability to maintain their balance while performing the 16 listed tasks. Score ranges from 0-100% and reflects overall % confidence. Lower scores indicate less confidence and thus worse outcome.
Parkinson's Disease Questionnaire Short Form | Prior to initiation of 8 week walking program and immediately upon completion
  Self-administered 8-question quality of life questionnaire for people with Parkinson disease, including 1 question from each of the following domains: mobility, ADLs, emotional well-being, stigma, social support, cognitions, communication, and bodily discomfort. Each question is scored 0-4 points and the scores are summed and divided by total possible to give a % score.
Trail Making Test A | Prior to initiation of 8 week walking program and immediately upon completion
  The Trail Making Test (TMT) is a test of visual conceptual and visuo-motor tracking that consists of two parts: Trail A and B. Trail A involves the individual connecting a sequence of 25 numbers distributed over a sheet of paper in order. Outcome measures for both tasks include time to completion (seconds).
Trail Making Test B | Prior to initiation of 8 week walking program and immediately upon completion
  The Trail Making Test (TMT) is a test of visual conceptual and visuo-motor tracking that consists of two parts: Trail A and B. Trail B requires the individual to alternately connect 25 numbers and letters (e.g. 1-A-2-B-3-C, etc). Outcome measures for both tasks include time to completion (seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Salido, DPT, PhD, Principal Investigator — Pacific Northwest University of Health Sciences
Locations (1):
- Pacific Northwest University of Health Sciences, Yakima, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warmerdam E, Romijnders R, Welzel J, Hansen C, Schmidt G, Maetzler W. Quantification of Arm Swing during Walking in Healthy Adults and Parkinson's Disease Patients: Wearable Sensor-Based Algorithm Development and Validation. Sensors (Basel). 2020 Oct 21;20(20):5963. doi: 10.3390/s20205963. PMID 33096899
- [Background] Shearin SM, McCain KJ, Querry R. Description of novel instrumented analysis of the Four Square Step Test with clinical application: A pilot study. Gait Posture. 2020 Oct;82:14-19. doi: 10.1016/j.gaitpost.2020.08.119. Epub 2020 Aug 20. PMID 32858317
- [Background] Salse-Batan J, Sanchez-Lastra MA, Suarez-Iglesias D, Varela S, Ayan C. Effects of Nordic walking in people with Parkinson's disease: A systematic review and meta-analysis. Health Soc Care Community. 2022 Sep;30(5):e1505-e1520. doi: 10.1111/hsc.13842. Epub 2022 May 20. PMID 35593147
- [Background] Cugusi L. Nordic Walking for the Management of People With Parkinson Disease: A Systematic Review - ClinicalKey. Accessed July 9, 2024. https://www-clinicalkey-com.proxy.pnwu.org/#!/content/playContent/1-s2.0-S1934148217302897?returnurl=null&referrer=null